CLINICAL TRIAL: NCT02418260
Title: Surgical Interventions for the Treatment of Humeral Shaft Fractures: Randomized Controlled Clinical Trial
Brief Title: Surgical Interventions for the Treatment of Humeral Shaft Fractures
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Rafael Pierami, Rafael Pierami, M.D., Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24997313.8.0000.5505
Record Dates: First submitted 2015-04-08; First posted 2015-04-16 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Fracture of Shaft of Humerus; Humerus Fracture
Keywords: Humerus; shaft; diaphyseal; fractures
MeSH Terms: conditions — Humeral Fractures; Fractures, Bone | interventions — Open Fracture Reduction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Open reduction and plate osteosynthesis (Active Comparator): Open reduction and internal fixation with DCP 4.5mm plate.
  Interventions: Procedure: Open reduction and plate osteosynthesis
- Bridge Plate (Experimental): Patients will be submitted to closed reduction and anterior bridge plate osteosynthesis (narrow 4.5mm DCP plate will be used)
  Interventions: Procedure: Bridge Plate osteosynthesis
- Intramedullary nail (Experimental): Patients will be submitted to closed reduction and locked intramedullary nail osteosynthesis.
  Interventions: Procedure: Locked intramedullary nail osteosynthesis

INTERVENTIONS:
Procedure: Bridge Plate osteosynthesis — Trough two anterior skin incisions, the 4.5mm narrow DCP plate will be placed on the anterior surface of the humerus and, after indirect reduction, it will be fixed to the bone with 2 proximal and 2 distal screws.
  Other Names: Bridge Plate
  Arms: Bridge Plate
Procedure: Locked intramedullary nail osteosynthesis — Trough an anterolateral approach to the shoulder, the supraspinatus tendon will be longitudinally splited allowing the insertion of the intramedullary nail.
  Other Names: IMN
  Arms: Intramedullary nail
Procedure: Open reduction and plate osteosynthesis — Trough an posterior or anterolateral approach, the fracture will be directly reduced and fixed with a broad DCP 4.5mm plate.
  Other Names: ORIF
  Arms: Open reduction and plate osteosynthesis

SUMMARY:
This study intends to determine the best surgical treatment for humeral shaft fractures. One third of the patients will be treated with open reduction and internal fixation with plate; one third, with bridge plate technique and the remaining third with locked intramedullary nail.

DETAILED DESCRIPTION:
Humerus diaphyseal fractures are amongst the most common of the appendicular skeleton. Despite the fact that the conservative treatment is still the gold standard for the majority of these fractures, this method was not proven to be superior when compared to the surgical treatment. Surgical options for the treatment of humeral shaft fractures range from open reduction and internal fixation with plate to minimally invasive methods (bridge plate and intramedullary nail) and the best method has yet to be determined. The goal of this study is to determine the best surgical option for the treatment of humeral shaft fractures. For this, will be recruited 105 patients with humeral shaft fractures, wich will be allocated, randomly, in 3 distinct groups. Each patient will be submitted to one of three possible methods of humerus osteosynthesis: open reduction and internal fixation with plate (ORIF), closed reduction and fixation with bridge plate or closed reduction and fixation with intramedullary nail. All data will be paired according to the age, gender, fracture classification, patient comorbidities and smoking habit. The Pearson's chi-square" test will be used to analyze the results of the three groups regarding categorical variables, and Student t-test (parametric) will be used to compare groups with respect to the numerical variables. The investigators expect to conclude that the methods of minimally invasive osteosynthesis of humeral shaft fractures have similar or better functional and radiographic outcomes, compared to the method of open reduction and internal fixation with a plate, with lesser risk of complications and an earlier return to activities.

ELIGIBILITY:
Inclusion Criteria:

* Complete fracture with angulation greater than 20 degrees, rotation greater than 30 degrees and/or shortening greater than 3 cm.
* Fractures located from 4 cm distal to the surgical neck to 2 cm proximal to the end of the medullary canal.

Exclusion Criteria:

* fractures older than 3 weeks
* pathologic fractures
* fractures with extension to elbow or shoulder joint
* patients with ipsilateral upper extremity fracture or injury
* fractures with associated neurologic injury
* patients with previous pathology of the shoulder, arm or elbow that cause pain or range of motion limitation
* patients who do not agree with the terms of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Changes in the Disabilities of the Arm, Shoulder and Hand (DASH) | 48 weeks
  The survey will be applied at 8, 24 and 48 weeks after the intervention

SECONDARY OUTCOMES:
Changes in the Visual Analog Scale for Pain (VAS) | 48 weeks
  The VAS survey will be applied 1, 8, 24 and 48 weeks after the intervention
Changes in the Constant-Murley Shoulder Outcome Score | 48 weeks
  The Score will be obtained at 8, 24 and 48 weeks after the intervention
Complications (nonunion, symptomatic malunion, hardware related issues, shoulder pain, infection, neurological injury and loss of range of motion of shoulder and/or elbow) | 48 weeks
  Complications are defined as nonunion, symptomatic malunion, hardware related issues, shoulder pain, infection, neurological injury and loss of range of motion of shoulder and/or elbow.
Radiographic angular deformity | at 48 weeks
  Radiographic angular residual deformity will be measured at 48 weeks after the surgical procedure.
Time to previous activities return | 48 weeks
  time to return to previous acitivities will bem described in weeks after the surgery
Failure (need for aditional surgical procedure) | 48 weeks
  Failure is described as need for aditional surgical procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Pierami, Principal Investigator — Federal University of São Paulo
Locations (1):
- Hand and Upper Limb Surgery Discipline, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] MANN RJ, NEAL EG. FRACTURES OF THE SHAFT OF THE HUMERUS IN ADULTS. South Med J. 1965 Mar;58:264-8. doi: 10.1097/00007611-196503000-00002. No abstract available. PMID 14261543
- [Background] Rose SH, Melton LJ 3rd, Morrey BF, Ilstrup DM, Riggs BL. Epidemiologic features of humeral fractures. Clin Orthop Relat Res. 1982 Aug;(168):24-30. PMID 7105548
- [Background] McKee MD LS. Humeral Shaft Fractures. Rockwood and Green's Fractures in Adults. 7th ed. Philadelphia: Lippincot Williams & Wilkins; 2009
- [Background] Baumgaertel F, Buhl M, Rahn BA. Fracture healing in biological plate osteosynthesis. Injury. 1998;29 Suppl 3:C3-6. doi: 10.1016/s0020-1383(98)95002-1. PMID 10341891
- [Background] Bhandari M, Guyatt GH, Swiontkowski MF. User's guide to the orthopaedic literature: how to use an article about a surgical therapy. J Bone Joint Surg Am. 2001 Jun;83(6):916-26. doi: 10.2106/00004623-200106000-00015. No abstract available. PMID 11407801
- [Background] Schulz KF, Altman DG, Moher D. CONSORT 2010 statement: Updated guidelines for reporting parallel group randomised trials. J Pharmacol Pharmacother. 2010 Jul;1(2):100-7. doi: 10.4103/0976-500X.72352. No abstract available. PMID 21350618
- [Background] Solway S, Beaton, D.E., McConnell, S., & Bombardier, C. The DASH Outcome measure user's manual (2nd Edition). Institute for Work & Health. Toronto2002.
- [Background] Orfale AG, Araujo PM, Ferraz MB, Natour J. Translation into Brazilian Portuguese, cultural adaptation and evaluation of the reliability of the Disabilities of the Arm, Shoulder and Hand Questionnaire. Braz J Med Biol Res. 2005 Feb;38(2):293-302. doi: 10.1590/s0100-879x2005000200018. Epub 2005 Feb 15. PMID 15785841
- [Background] Flandry F, Hunt JP, Terry GC, Hughston JC. Analysis of subjective knee complaints using visual analog scales. Am J Sports Med. 1991 Mar-Apr;19(2):112-8. doi: 10.1177/036354659101900204. PMID 2039061
- [Background] Constant CR, Murley AH. A clinical method of functional assessment of the shoulder. Clin Orthop Relat Res. 1987 Jan;(214):160-4. PMID 3791738
- [Result] Balfour GW, Marrero CE. Fracture brace for the treatment of humerus shaft fractures caused by gunshot wounds. Orthop Clin North Am. 1995 Jan;26(1):55-63. PMID 7838503
- [Result] Sarmiento A, Kinman PB, Galvin EG, Schmitt RH, Phillips JG. Functional bracing of fractures of the shaft of the humerus. J Bone Joint Surg Am. 1977 Jul;59(5):596-601. PMID 873955
- [Result] Ward EF SF, Hughes JL. Fractures of the diaphyseal humerus. In: Saunders, ed. Skeletal trauma: fractures, dislocation, ligamentous injuries. Philadelphia: Saunders; 1998:1523-47
- [Result] Balfour GW, Mooney V, Ashby ME. Diaphyseal fractures of the humerus treated with a ready-made fracture brace. J Bone Joint Surg Am. 1982 Jan;64(1):11-3. No abstract available. PMID 7054192
- [Result] Amillo S, Barrios RH, Martinez-Peric R, Losada JI. Surgical treatment of the radial nerve lesions associated with fractures of the humerus. J Orthop Trauma. 1993;7(3):211-5. doi: 10.1097/00005131-199306000-00002. PMID 8326423
- [Result] Foster RJ, Swiontkowski MF, Bach AW, Sack JT. Radial nerve palsy caused by open humeral shaft fractures. J Hand Surg Am. 1993 Jan;18(1):121-4. doi: 10.1016/0363-5023(93)90255-2. PMID 8423295
- [Result] Pollock FH, Drake D, Bovill EG, Day L, Trafton PG. Treatment of radial neuropathy associated with fractures of the humerus. J Bone Joint Surg Am. 1981 Feb;63(2):239-43. PMID 7462281
- [Result] Ekholm R, Tidermark J, Tornkvist H, Adami J, Ponzer S. Outcome after closed functional treatment of humeral shaft fractures. J Orthop Trauma. 2006 Oct;20(9):591-6. doi: 10.1097/01.bot.0000246466.01287.04. PMID 17088659
- [Result] Rutgers M, Ring D. Treatment of diaphyseal fractures of the humerus using a functional brace. J Orthop Trauma. 2006 Oct;20(9):597-601. doi: 10.1097/01.bot.0000249423.48074.82. PMID 17088660
- [Result] Jawa A, McCarty P, Doornberg J, Harris M, Ring D. Extra-articular distal-third diaphyseal fractures of the humerus. A comparison of functional bracing and plate fixation. J Bone Joint Surg Am. 2006 Nov;88(11):2343-7. doi: 10.2106/JBJS.F.00334. PMID 17079389
- [Result] Gosler MW, Testroote M, Morrenhof JW, Janzing HM. Surgical versus non-surgical interventions for treating humeral shaft fractures in adults. Cochrane Database Syst Rev. 2012 Jan 18;1(1):CD008832. doi: 10.1002/14651858.CD008832.pub2. PMID 22258990
- [Result] Papasoulis E, Drosos GI, Ververidis AN, Verettas DA. Functional bracing of humeral shaft fractures. A review of clinical studies. Injury. 2010 Jul;41(7):e21-27. doi: 10.1016/j.injury.2009.05.004. Epub 2009 Jun 11. PMID 19523625
- [Result] Zagorski JB, Latta LL, Zych GA, Finnieston AR. Diaphyseal fractures of the humerus. Treatment with prefabricated braces. J Bone Joint Surg Am. 1988 Apr;70(4):607-10. PMID 3356728
- [Result] Wallny T, Westermann K, Sagebiel C, Reimer M, Wagner UA. Functional treatment of humeral shaft fractures: indications and results. J Orthop Trauma. 1997 May;11(4):283-7. doi: 10.1097/00005131-199705000-00011. PMID 9258827
- [Result] Fjalestad T, Stromsoe K, Salvesen P, Rostad B. Functional results of braced humeral diaphyseal fractures: why do 38% lose external rotation of the shoulder? Arch Orthop Trauma Surg. 2000;120(5-6):281-5. doi: 10.1007/s004020050465. PMID 10853896
- [Result] Koch PP, Gross DF, Gerber C. The results of functional (Sarmiento) bracing of humeral shaft fractures. J Shoulder Elbow Surg. 2002 Mar-Apr;11(2):143-50. doi: 10.1067/mse.2002.121634. PMID 11988725
- [Result] Ricciardi-Pollini PT, Falez F. The treatment of diaphyseal fractures by functional bracing. Results in 36 cases. Ital J Orthop Traumatol. 1985 Jun;11(2):199-205. PMID 4066292
- [Result] Persad IJ, Kommu S. U cast or functional bracing following fractures of the shaft of humerus. Emerg Med J. 2007 May;24(5):361. doi: 10.1136/emj.2007.048504. No abstract available. PMID 17452711
- [Result] Wallny T, Sagebiel C, Westerman K, Wagner UA, Reimer M. Comparative results of bracing and interlocking nailing in the treatment of humeral shaft fractures. Int Orthop. 1997;21(6):374-9. doi: 10.1007/s002640050189. PMID 9498146
- [Result] Bell MJ, Beauchamp CG, Kellam JK, McMurtry RY. The results of plating humeral shaft fractures in patients with multiple injuries. The Sunnybrook experience. J Bone Joint Surg Br. 1985 Mar;67(2):293-6. doi: 10.1302/0301-620X.67B2.3980544.
- [Result] Dabezies EJ, Banta CJ 2nd, Murphy CP, d'Ambrosia RD. Plate fixation of the humeral shaft for acute fractures, with and without radial nerve injuries. J Orthop Trauma. 1992;6(1):10-3. PMID 1556609
- [Result] Heim D, Herkert F, Hess P, Regazzoni P. Surgical treatment of humeral shaft fractures--the Basel experience. J Trauma. 1993 Aug;35(2):226-32. PMID 8355300
- [Result] Grass G, Kabir K, Ohse J, Rangger C, Besch L, Mathiak G. Primary Exploration of Radial Nerve is Not Required for Radial Nerve Palsy while Treating Humerus Shaft Fractures with Unreamed Humerus Nails (UHN). Open Orthop J. 2011;5:319-23. doi: 10.2174/1874325001105010319. Epub 2011 Aug 26. PMID 21915231
- [Result] Chao TC, Chou WY, Chung JC, Hsu CJ. Humeral shaft fractures treated by dynamic compression plates, Ender nails and interlocking nails. Int Orthop. 2005 Apr;29(2):88-91. doi: 10.1007/s00264-004-0620-8. Epub 2005 Feb 16. PMID 15714304
- [Result] Ajmal M, O'Sullivan M, McCabe J, Curtin W. Antegrade locked intramedullary nailing in humeral shaft fractures. Injury. 2001 Nov;32(9):692-4. doi: 10.1016/s0020-1383(01)00076-6. PMID 11600115
- [Result] Petsatodes G, Karataglis D, Papadopoulos P, Christoforides J, Gigis J, Pournaras J. Antegrade interlocking nailing of humeral shaft fractures. J Orthop Sci. 2004;9(3):247-52. doi: 10.1007/s00776-004-0780-9. PMID 15168178
- [Result] Aksu N, Karaca S, Kara AN, Isiklar ZU. Minimally invasive plate osteosynthesis (MIPO) in diaphyseal humerus and proximal humerus fractures. Acta Orthop Traumatol Turc. 2012;46(3):154-60. doi: 10.3944/aott.2012.2592. PMID 22659630
- [Result] Shetty MS, Kumar MA, Sujay K, Kini AR, Kanthi KG. Minimally invasive plate osteosynthesis for humerus diaphyseal fractures. Indian J Orthop. 2011 Nov;45(6):520-6. doi: 10.4103/0019-5413.87123. PMID 22144745
- [Result] Ouyang H, Xiong J, Xiang P, Cui Z, Chen L, Yu B. Plate versus intramedullary nail fixation in the treatment of humeral shaft fractures: an updated meta-analysis. J Shoulder Elbow Surg. 2013 Mar;22(3):387-95. doi: 10.1016/j.jse.2012.06.007. Epub 2012 Sep 1. PMID 22947239
- [Result] Liu GD, Zhang QG, Ou S, Zhou LS, Fei J, Chen HW, Nan GX, Gu JW. Meta-analysis of the outcomes of intramedullary nailing and plate fixation of humeral shaft fractures. Int J Surg. 2013;11(9):864-8. doi: 10.1016/j.ijsu.2013.08.002. Epub 2013 Aug 28. PMID 23994004
- [Result] Wang X, Chen Z, Shao Y, Ma Y, Fu D, Xia Q. A meta-analysis of plate fixation versus intramedullary nailing for humeral shaft fractures. J Orthop Sci. 2013 May;18(3):388-97. doi: 10.1007/s00776-013-0355-8. Epub 2013 Mar 8. PMID 23471713
- [Result] Bhandari M, Devereaux PJ, McKee MD, Schemitsch EH. Compression plating versus intramedullary nailing of humeral shaft fractures--a meta-analysis. Acta Orthop. 2006 Apr;77(2):279-84. doi: 10.1080/17453670610046037. PMID 16752291
- [Result] Kurup H, Hossain M, Andrew JG. Dynamic compression plating versus locked intramedullary nailing for humeral shaft fractures in adults. Cochrane Database Syst Rev. 2011 Jun 15;2011(6):CD005959. doi: 10.1002/14651858.CD005959.pub2. PMID 21678350